CLINICAL TRIAL: NCT02161172
Title: Cognitive, Functional, and Psychosocial Outcome After Mild Traumatic Brain Injury: a Cross-sectional Study at a Tertiary Care Trauma Center.
Brief Title: Cognitive and Psychosocial Outcome After Mild Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Chen, Doctor, Shanghai 6th People's Hospital
Other Study IDs: 658214
Record Dates: First submitted 2014-06-10; First posted 2014-06-11 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Mild traumatic brain injury; Cognitive outcome; Psychological outcome
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mild traumatic brain injury: Traumatic brain injury patients with Glasgow coma score (GCS) of 13-15.

SUMMARY:
Patients with traumatic brain injury are likely to present with cognitive, psychological, emotional and behavioral problems during different periods, all of which affect patients' life quality seriously. The aim of this study was to assess cognitive and psychosocial outcome in patients with mild traumatic brain injury, and to determine the risk factors associated with cognitive and psychological outcome. Mini-mental state examination (MMSE), activities of daily living scale (ADL), the Hospital Anxiety Depression Scale (HADS) and mental health symptom checklist (SCL-90) were used to assess the cognitive performance and psychological outcomes in 360 patients with mild traumatic brain injury. Chi-square, Fisher's exact tests and Logistic regression analysis were used to analyze the risk factors.

ELIGIBILITY:
Inclusion Criteria:

* 18 ~ 60 years old
* Education: primary school and above, who could understand the content of psychological test
* History of brain trauma
* No taking of antipsychotic or any other drugs affecting central nervous system before the test
* Glasgow coma score (GCS) was 13-15

Exclusion Criteria:

* History of craniocerebral injury, brain disease, mental disease
* With mental retardation
* with other serious body diseases
* History of drug and alcohol dependence
* With color-blind or color weakness
* Who had severe visual and auditory disorders after brain injury
* Who failed or failed in completing the test effectively
* With cognitive impairment caused by the damage of the unilateral frontal or bilateral lobes, or with language dysfunction caused by temporal lobe damage

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 360 patients with mild traumatic brain injury were enrolled in this study. Their age ranged from 18 to 60 years, with mean age of 54.3 years. Types of trauma included scalp hematoma, scalp laceration, cerebral contusion, subarachnoid hemorrhage, cerebral concussion, epidural hematoma, subdural hematoma and skull fracture. Mechanisms of injury contained traffic accident, fall, industrial accident, etc. Occupation of patients included cadres, workers, farmers, individual, unemployed. Education: college or above, middle school, primary school.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination | 6 months
  MMSE includes seven factors, namely: the time orientation factor (5 points), place orientation (5 points), immediate memory (3 points), short-term memory (3 points), calculation capabilities (5 points), verbal expression, naming and repetition (4 points), speech reading and understanding (4 points), graphic depiction (1 points). The scales for the description of cognitive function impairment were grouped into three levels of education: illiteracy (17 points), primary school (20 points) and middle school (24 points). The one with score below average was considered with cognitive function impairment.

SECONDARY OUTCOMES:
Activity of daily living scale | 6 months
  The scale is divided into two parts: physical self-care ability, instrumental activities of daily living. 1 point for each option means normal; If 2~4 points for one option, he or she probably had ability decline; If two or more parts ≥3 points or total score≥ 22 points (14 questions), he or she exhibited living ability decline clearly.

OTHER OUTCOMES:
Hospital anxiety and depression Scale | 6 months
  The scale includes 14 items and each has 0-3 points. The score of the former seven items > 7, indicating depression symptom; the later seven items > 7, indicating anxiety symptom.
Symptom Check-List 90 | 6 months
  This scale has been widely used to patients with neurosis, adjustment disorder and other slight mental psychological disorder. According to the national norm results, if the total score > 160, or the number of positive items > 43, or one factor score >2, we consider the positive screening.

CONTACTS AND LOCATIONS:
Overall Officials: Heng-Li Tian, M.D., Ph.D., Study Director — Shanghai 6th People's Hospital
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, China